CLINICAL TRIAL: NCT06937801
Title: A Randomized, Double-blind, Placebo-controlled Clinical Trial to Assess the Effect of Collagen Peptide on Perceived Gastrointestinal Discomfort in Healthy Adult Participants With Presence of Gastrointestinal Symptoms
Brief Title: To Assess the Effect of Collagen on Gastrointestinal Discomfort in Healthy Adults With Gastrointestinal Symptoms.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rousselot BVBA (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R02-24-01-T0070
Record Dates: First submitted 2025-04-04; First posted 2025-04-22 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Gastrointestinal Disorders
Keywords: Gastrointestinal discomfort; gastrointestinal symptoms
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): single dose
  Interventions: Other: Placebo
- Collagen Peptide (Active Comparator): Dissolve in water, single dose, 10 g
  Interventions: Dietary Supplement: Collagen Peptide

INTERVENTIONS:
Dietary Supplement: Collagen Peptide — 10g Collagen Hydrolysate per sachet
  Arms: Collagen Peptide
Other: Placebo — Placebo - active ingredients: N/A
  Arms: Placebo

SUMMARY:
This study will enroll healthy adults with perceived gastrointestinal symptoms to evaluate the effect of collagen peptides compared to placebo.

DETAILED DESCRIPTION:
This double-blind, placebo-controlled trial aims to assess the efficacy of collagen peptides in addressing gastrointestinal discomfort, gut microbiota composition, gut permeability, mood, anxiety, perceived stress, quality of life and cognitive function. The study will include healthy adults experiencing gastrointestinal symptoms while excluding individuals with chronic illnesses or recent infections that might impact the results.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults from 18 to 64 years of age (inclusive).
2. Have a BMI between 18.0 to 34.9 kg/m2 (inclusive).
3. In good general health as determined by the investigator.
4. Are able to consume an animal-sourced powder product when mixed with water and taken orally.
5. Have a presence of GI symptoms as confirmed by a GSRS average score between 2 and 5 (inclusive).
6. Have maintained consistent dietary habits, including medication and supplement intake, and lifestyle for the last 3 months before screening and agree to maintain them throughout the study.
7. Agree to avoid anal penetration for 72 h prior to each fecal sample collection.
8. Agree to follow the restrictions on concomitant treatments, and lifestyle.
9. Agree to follow the restrictions on lifestyle.
10. Agree to use acceptable contraceptive methods.
11. Willing and able to give voluntary consent, able to understand and read the questionnaires, carry out all study-related procedures and agree to the requirements of this study.

Exclusion Criteria:

1. Individuals who are lactating, pregnant or planning to become pregnant during the study.
2. Have a known sensitivity, intolerability, or allergy to any of the study products or their excipients.
3. Current COVID-19 infections, or currently have the post COVID-19 condition as defined by World Health Organization (WHO).
4. Recent history of an episode of acute GI illness such as nausea, vomiting, or diarrhea.
5. Have Type I diabetes, uncontrolled Type II diabetes, uncontrolled high blood pressure (≥140 systolic or ≥90 diastolic mmHg), or uncontrolled thyroid disease ("uncontrolled" defined as being unmedicated, have an unstable use of medication within 3 months prior to screening, or have a stable use of medication for 3 months but still have uncontrolled conditions).
6. Have a current diagnosis or history of irritable bowel syndrome (IBS), inflammatory bowel disease (IBD), functional constipation or diarrhea (defined by the ROME IV diagnostic criteria), celiac disease, malabsorption, gastroparesis, endometriosis or eating disorder.
7. Have a chronic inflammatory condition/disease (e.g., rheumatoid arthritis, ulcerative colitis, lupus).
8. Have medical condition(s) known to interfere with absorption, distribution, metabolism, or excretion of the study product (e.g., Crohn's disease, short bowel, acute or chronic pancreatitis, or pancreatic insufficiency).
9. Have a history of heart/cardiovascular disease, renal disease (dialysis or renal failure), hepatic impairment/disease, immune disorders and/or immunocompromised (i.e., HIV/AIDS).
10. Have a history of cancer (except localized skin cancer without metastases or in situ cervical cancer), unless recovery occurred more than 5 years before the screening visit.
11. Are receiving treatments for or have been hospitalized in the last 12 months for psychiatric disorders (e.g., depression, generalized anxiety disorder, bipolar disorder, schizophrenia, etc.).
12. Reports a clinically significant illness during the 28 days before the first dose of study product.
13. Major surgery in 3 months prior to screening or planned major surgery during the study.
14. Have a history of alcohol or substance abuse in the 12 months prior to screening (including having been hospitalized for such in an in-patient or out-patient intervention program) or use that in the opinion of the investigator may be of a concern for the study.
15. Current enrollment or past participation in another study with any product(s) with at least one active ingredient within 28 days before first dose of study product or longer.
16. Living in the same household as another currently/previously enrolled participant in the present study.
17. Any other medical condition/situation or use of medications/supplements/therapies that, in the opinion of the investigator, may adversely affect the participant's ability to participate in the study or its measures or pose a significant risk to the participant.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2025-05-08 (Actual); Primary Completion 2025-11-21 (Actual); Study Completion 2025-11-21 (Actual)

PRIMARY OUTCOMES:
To assess the impact of the Test Product on perceived GI discomfort in healthy adults compared to a placebo | Baseline to Week 8
  Gastrointestinal Symptom Rating Scale (GSRS) total score (From 1-7). A higher score is a worse outcome.

SECONDARY OUTCOMES:
To assess the impact of the TP on perceived GI symptoms in healthy adults compared to a placebo | Baseline to Week 8
  GSRS dimension scores of reflux, diarrhea, abdominal pain, indigestion and constipation. Score (From 1-7). A higher score is a worse outcome.
To assess the impact of the TP on perceived GI discomfort and symptoms in healthy adults compared to a placebo | Baseline to Week 4
  GSRS total score and dimension scores of reflux, diarrhea, abdominal pain, indigestion and constipation. Score (From 1-7). A higher score is a worse outcome.
To assess the effect of the TP on the modulation of the gut microbiota composition, in particular growth stimulation of beneficial bacteria, in healthy adults compared to a placebo | Baseline to Week 8
  Change in the abundance of Bifidobacteriaceae (B. longum) in the stool sample as assessed by qPCR
To assess the effect of the TP on the modulation of the gut microbiota composition, in particular growth stimulation of beneficial bacteria, in healthy adults compared to a placebo | Baseline to Week 8
  Change in the abundance of Bifidobacteriaceae (B. bifidum) in the stool sample as assessed by qPCR
To assess the effect of the TP on the modulation of the gut microbiota composition, in particular growth stimulation of beneficial bacteria, in healthy adults compared to a placebo | Baseline to Week 8
  Change in the abundance of Pevotellaceae (P. copri) in the stool sample as assessed by qPCR
To assess the effect of the TP on the modulation of the gut microbiota composition, in particular growth stimulation of beneficial bacteria, in healthy adults compared to a placebo | Baseline to Week 8
  Change in the abundance of Pevotellaceae (P. Stercorea) in the stool sample as assessed by qPCR
To assess the effect of the TP on the modulation of the gut microbiota composition, in particular growth stimulation of beneficial bacteria, in healthy adults compared to a placebo | Baseline to Week 8
  Change in the abundance of Bacteroides (B. Cellulosilyticus) in the stool sample as assessed by qPCR
To assess the effect of the TP on the modulation of the gut microbiota composition, in particular growth stimulation of beneficial bacteria, in healthy adults compared to a placebo | Baseline to Week 8
  Change in the abundance of Bacteroides (B. thetaiotaomicron) in the stool sample as assessed by qPCR
To assess the effect of the TP on the modulation of the gut microbiota composition, in particular growth stimulation of beneficial bacteria, in healthy adults compared to a placebo | Baseline to Week 8
  Change in the abundance of Bacteroides (B. intestinalis) in the stool sample as assessed by qPCR
To assess the effect of the TP on the modulation of the gut microbiota composition, in particular growth stimulation of beneficial bacteria, in healthy adults compared to a placebo | Baseline to Week 8
  Change in the abundance of Bacteroides (B. caecimuris) in the stool sample as assessed by qPCR
To assess the effect of the TP on the modulation of the gut microbiota composition, in particular growth stimulation of beneficial bacteria, in healthy adults compared to a placebo | Baseline to Week 8
  Change in the abundance of Bacteroides (B. fragilis) in the stool sample as assessed by qPCR
To assess the effect of the TP on the modulation of the gut microbiota composition, in particular growth stimulation of beneficial bacteria, in healthy adults compared to a placebo | Baseline to Week 8
  Change in the abundance of Lactobacillaceae (L. salivarus) in the stool sample as assessed by qPCR
To assess the effect of the TP on the modulation of the gut microbiota composition, in particular growth stimulation of beneficial bacteria, in healthy adults compared to a placebo | Baseline to Week 8
  Change in the abundance of Lactobacillaceae (L. paracasei) in the stool sample as assessed by qPCR
To assess the effect of the TP on the modulation of the gut microbiota composition, in particular growth stimulation of beneficial bacteria, in healthy adults compared to a placebo | Baseline to Week 8
  Change in the abundance of Ruminococccaceae (F. prausnitzii) in the stool sample as assessed by qPCR
To assess the effect of the TP on the modulation of the gut microbiota composition, in particular growth stimulation of beneficial bacteria, in healthy adults compared to a placebo | Baseline To Week 8
  Change in the abundance of Lachnospiraceae (R. hominis) in the stool sample as assessed by qPCR.
To assess the effect of the TP on mood/anxiety in healthy adults compared to a placebo | Baseline to Week 8
  Change in Brunnel Mood Scale questionnaire scores or anger, confusion, depression, fatigue, tension and vigour. The Scale is from 0-16, a higher score is worse.
To assess the effect of the TP on perceived stress in healthy adults compared to a placebo | Baseline to Week 8
  Change in Perceived Stress Scale -10 score - The score is from 0-40, a higher score is worse.
To assess the effect of the TP on quality of life in healthy adults compared to a placebo | Baseline to Week 8
  Change in Research and Development Short Form - 36 score. The score is from 0-100, a higher score is better.
To assess the effect of the TP on cognitive function in healthy adults compared to a placebo | Baseline to Week 8
  Change from baseline to Week 8 in Trail Making Test score. Time is recorded in seconds to complete the test, a higher time is worse.
To assess the effect of the TP on cognitive function in healthy adults compared to a placebo | Week 8
  Change in Dimensional Change Card Sort Test score of executive function. The score is from 0-12, a higher score is better..
To assess the effect of the TP on cognitive function in healthy adults compared to a placebo | Baseline to Week 8
  Change in Flanker Inhibitory Control and Attention Test score of executive function. The test measures time in milliseconds, a higher time is worse.
To assess the effect of the TP on cognitive function in healthy adults compared to a placebo | Baseline to Week 8
  Change in Stroop Colour and Word Test score of executive function. The test measures time in milliseconds, a higher time is worse.
To assess the effect of the TP on intestinal permeability in healthy adults compared to a placebo | Baseline to Week 8
  Change in serum LPS levels

OTHER OUTCOMES:
To assess the safety of the TP | Baseline to Week 8
  Vital Signs : Heart rate (beats per minute)
To assess the safety of the TP | Baseline to Week 8
  Vital Signs: Blood pressure (mmhg)
To assess the safety of the TP | Baseline to Week 8
  Anthropometrics: Weight (kilograms)
To assess the safety of the TP | Baseline to Week 8
  Anthropometrics: BMI (Body Mass Index) in body weight (kilograms) divided by the square of their height (meters)
To assess the safety of the TP | Baseline to Week 8
  Report Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Nicoletta Virgilio, Study Director — Rousselot BV
Locations (1):
- Nutrasource Site (Apex Trials), Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No